CLINICAL TRIAL: NCT02255578
Title: Phase 3 Study Investigating the Effect of Endobarrier Treatment on Fertility in Women With Polycystic Ovary Syndrome
Brief Title: Endobarrier Treatment in Women With PCOS
Acronym: EPCOS
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Gabriella Segal-Lieberman, Endocrinologist, Sheba Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHEBA-14-1170-GL-CTIL
Record Dates: First submitted 2014-07-09; First posted 2014-10-02 (Estimated); Last update posted 2014-10-02 (Estimated); Status verified 2014-09

CONDITIONS: Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- IVF treatment (Other): Fertility, as determined by egg quality parameters, as well as metabolic parameters, will be assessed following Endobarrier treatment in PCOS during IVF treatment.
  Interventions: Device: Endobarrier treatment in PCOS
- clomiphene citrate treatment (Other): Ovulation rate in response to clomiphen citrate after Endobarrier treatment in PCOS.
  Interventions: Device: Endobarrier treatment in PCOS; Drug: clomiphene citrate treatment

INTERVENTIONS:
Device: Endobarrier treatment in PCOS — the effect of an EndoBarrier device on fertility and metabolic parameters in obese insulin resistant (IR) PCOS women
Drug: clomiphene citrate treatment
  Arms: clomiphene citrate treatment

SUMMARY:
Women with Polycystic ovary syndrome (PCOS) experience multiple fertility treatments, a long treatment duration and a low pregnancy prevalence. This syndrome is frequently accompanied by overweight and insulin resistance which can mediate the limited response to fertility treatment. The Endobarrier device was shown to be efficient in weight and glucose lowering. The aim of this study is to investigate the ability of the Endobarrier device to improve the outcome of fertility treatments in women with PCOS.

DETAILED DESCRIPTION:
1. PCOS Polycystic ovary syndrome (PCOS) is the most common endocrinopathy among women of reproductive age, associated with reproductive and metabolic dysfunction with a prevalence of 5-10% of reproductive aged women.

   Diagnostic criteria vary and according to the Rotterdam ESHRE/ASRM- Sponsored PCOS Consensus Workshop Group PCOS is defined when at least two of the following three criteria are present: [i] polycystic ovaries, by ultrasound [ii] oligo and/or anovulation, and [iii] clinical and/or biochemical signs of hyperandrogenism.

   The clinical presentation varies from amenorrhea and a sonographic picture of polycystic ovaries but with subtle phenotypic abnormalities or signs of hyperandrogenism, to advanced Stein and Leventhal syndrome with clinical heterogeneity as the rule. Moreover, women with PCOS might exhibit features of the metabolic syndrome, including impaired glucose tolerance (IGT), obesity and dyslipidaemia ,with their associated long- term sequelae, namely endometrial carcinoma, hypertension, type 2 diabetes (T2D) and cardiovascular disease.

   Impaired Glucose Intolerance (IGT) and PCOS Impaired glucose tolerance, or insulin resistance, are defined as decreased insulin-mediated glucose utilization. It has long been recognized as a major risk factor for diabetes. Moreover, it was shown that lifestyle intervention or metformin in patients with IGT, may reduce the prevalence of T2D. Several dynamic invasive tests and calculated indices are currently available for detecting IGT. While the euglycemic clamp technique is considered the most accurate test for the assessment of insulin resistance, this cumbersome test is frequently replaced by the simple measurement of the ratio of fasting glucose to fasting insulin, or the 2-hour glucose level after a 75-g oral glucose tolerance test (OGTT) (WHO criteria, impaired glucose tolerance [IGT] >140 mg/dL to 199 mg/dL). As a result, reports of the prevalence on IGT in women with PCOS vary depending on the sensitivity and specificity of the tests employed and the heterogenic phenotypes of PCOS.

   Obesity - definition, significance and prevalence among women with PCOS:

   Obesity, a common clinical manifestation of PCOS patients, is linked to insulin resistance and failure or delayed response to the various COH treatments.The associated health detriments of this major health problem are increased with increasing body mass index (BMI). Data regarding the impact of obesity on IVF cycles outcome is controversial, ranging from studies reporting on no effect of increasing BMI on IVF success rates to those demonstrating a lower cumulative live birth rates in overweight patients. PCOS and assisted reproduction PCOS women with insulin resistance undergoing ovulation induction with gonadotropin have a longer duration of treatment, use a higher total FSH dose, have an elevated cancellation rate and a lower conception rate. Improving insulin sensitivity through both lifestyle and pharmacological intervention were suggested to ameliorate the aforementioned abnormalities, restore ovulation and enhance pregnancy in women with PCOS.

   In vitro fertilization (IVF) and embryo transfer (ET) is an effective therapy for PCOS patients and results in pregnancy rates that are comparable with those for women with tubal factor infertility. Moreover, because the number of multiple pregnancies can be kept to a minimum by transferring small numbers of embryos, IVF-ET became a reasonable option to PCOS patients who are refractory to conventional infertility modalities or who have coexisting infertility factors.

   Many controlled ovarian hyperstimulation (COH) strategies have been offered for the treatment of patients with PCOS undergoing IVF.

   In an attempt to examine the influence of BMI on IVF outcome in patients undergoing COH with either GnRH-agonist or antagonist, the investigators found that while in patients with BMI>25 kg/m2, COH with either GnRH-agonist or antagonist achieved a comparable outcome, in those with BMI<25 kg/m2, the use of GnRH-agonist suppressive protocol revealed a significantly higher pregnancy rates.

   Moreover, in another study of PCOS patients undergoing IVF-ET cycles, the investigators demonstrated that COH utilizing the midluteal long GnRH-agonist suppressive protocol was the protocol of choice in lean patients, probably due to its ability to lower the high basal LH milieu and its detrimental effect of oocytes' quality and implantation potential.
2. Device Description ENDOBARRIER The EndoBarrier Gastrointestinal Liner system received CE Mark on 11 December 2009 and is indicated for the treatment of obesity and Type 2 diabetes. The implant is indicated for a maximum implant duration period of twelve months. The intent of the EndoBarrier is to facilitate glycemic control and weight loss by mimicking portions of the Roux-en-Y bypass procedure. The device consists of 3 components: the implant, the delivery system, and the removal system.

The procedure entails bypassing the duodenum and the proximal jejunum with a 60 cm non-permeable polymeric sleeve which is attached to the duodenal wall. This sleeve prevents the contact of food with the duodenal wall, thereby re-capitulating one of the major properties of the RYGB operation. With this technique, control of diabetes is accompanied by weight loss, with no need for medications that may cause weight gain / hypoglycemia and may serve to replace or postpone surgery.

In a recent paper by de Moura et al, Twenty-two subjects with uncontrolled type 2 diabetes and a body mass index between 40- 60 kg/m ² were implanted with the EndoBarrier and followed prospectively for 1 year.

The authors found statistically significant reductions in fasting blood glucose (- 30.3 ± 10.2 mg/dL), fasting insulin (- 7.3 ± 2.6 lU/mL), and HbA1c ( - 2.1±0.3%) in patients undergoing the procedure.

The study conclusions were that EndoBarrier improves glycemic status in obese subjects with diabetes and therefore represents a non-surgical, reversible alternative to bariatric surgery. Internal data from GI Dynamics reveals that obese subject (average BMI of 44 kg/m²) and uncontrolled diabetes ( average A1c of 8.4 %) who were implanted with EndoBarrier for one year showed the following:

1. A reduction of 2.1% of the A1c level, with a value of less than 7% in 80% of the subjects.
2. An average reduction of 20 Kg (representing 16% of the excess weight).
3. A 29% reduction in the triglyceride level and a 14% reduction in LDL-c. After 12 months the EndoBarrier was removed and the subjects remained in follow up for additional 18 months. During this period, the achievement was maintained.

3. Study Design: This is a two arm open-label three phase trail investigating the effect of an EndoBarrier device on fertility and metabolic parameters in obese insulin resistant (IR) PCOS women Arm 1: women seeking pregnancy after failed IVF treatment cycle/s. Arm 2: women seeking pregnancy after failure to ovulate in response to clomiphene citrate (CC) - clomiphene resistant.

Phase 1: (treatment phase) - Six months with Endobarrier Phase 2: (follow-up phase) - Twelve months after Endobarrier retrieval Phase 3: (long term observation phase) - to see whether and when a pregnancy was achieved within the second year after retrieval.

4. Methods and assessments: 4.1 Visit 1- screening All potential patients will be screened for eligibility at visit 1. Informed consent (ICF) will be explained to the patient prior to conducting any study procedures. A discussion in which the patient is explained about the advantage and disadvantage of the trail and the trail procedures will be taken. If participation is agreed to by the patient after they read the ICF, the patient will sign and date the ICF, and get a copy of the signed and dated form.

The following activities will occur on Visit 1:

The patient signs the ICF form A patient number will be assigned to the patient. Inclusion / Exclusion criteria will be reviewed. Demographic data : Age. Medical history evaluation and concomitant medication record. A physical and gynecological examination (including Ultrasound of Ovaries) will be conducted.

An oral OGTT 75g will be performed. Fasting Laboratory measurements will be performed A date for visit 2 will be scheduled.

4.2 visit 2 - Gastro screening

The following activities will occur on Visit 2:

The patient will be referred to the Gastroenterology department for Gastroscopy.

The patient will be instructed to start 40 mg Omeprazole twice daily 3 days prior to visit 4 (Implantation of the Endobarrier).

The patient will be instructed to start contraceptive from now on. Diet consultation will be performed The patient will be asked to answer the "Visual analog scale" (VAS) questionnaire.

A date for visit 3 will be scheduled.

4.3 visit 3 - Endobarrier implantation The patient will arrive in a fasting state. The patient will be asked about any AE's and change in medications. Vital signs, weight, waist circumferences will be measured. Fasting Laboratory measurements will be performed Under full anesthesia (in order to achieve the best conditions for the accurate positioning of the device) gastroscopy will be performed and a guide wire will be inserted to the jejunum.

The Endobarrirer device will be inserted over the guide wire and introduced into the duodenal bulb. The correct location of the device will be evaluated by the endoscope.

Under fluoroscopy the device will be operated and the sleeve will be released from its capsule. Contrast material will be injected thorough the sleeve to insure full opening.

After full expansion of the sleeve, the anchoring mechanism will be operated and the sleeve will be anchored by small hooks to the duodenal bulb.

Correct hooking will be visualized endoscopically.

4.4 visits 4-9 The patient will be asked about any AE's and change in medications. Vital signs, weight, waist circumferences will be measured. Fasting Laboratory measurements will be performed Diet consultation will be performed. The patient will be asked to answer the "Visual analog scale" (VAS) questionnaire.

4.5 visit 10- pre-retrieval visit The patient will be asked about any AE's and change in medications. Vital signs, weight, waist circumferences will be measured. Fasting laboratory measurements will be performed The patient will be asked to answer the "Visual analog scale" (VAS) questionnaire

4.6 visit 11- Endobarrier retrieval The retrieval procedure will be performed after sedation. A retrieval hood will be connected to the endoscope tip. A scope will be introduced to the duodenum. A retrieval grasper will be inserted through the scope. By pulling the drawstring the anchoring hook will collapse and when all hooks are within the plastic retrieval hood the endoscope will be withdrawn safely out.

The patients will be referred to the infertility Clinic for treatment.

4.7 visit 12-19 - once in 3M follow up Patient will come to a visit once every 3 months, until pregnancy is achieved or until the end of the study period.

Patient will be asked about any AE's and change in medications. Gynecological exam (may include Ultrasound of Ovaries) may be performed. Fasting laboratory measurements will be performed The patient will be asked to answer the "Visual analog scale" (VAS) questionnaire.

Patient will be required to provide the site will data regarding last fertility treatment

**In case pregnancy is achieved patient is requested to inform the site within 1 week.

Relevant information regarding the fertility treatment will be collected

ELIGIBILITY:
Inclusion criteria:

1. Women willing to comply with study requirements and have signed an informed consent form.
2. Age 20-35
3. BMI ≥ 35 kg/m²
4. A history of failed IVF treatment cycle/s or resistance to ovulation induction with clomiphene citrate.
5. Documented negative pregnancy test.
6. Women agree to remain on contraceptives as long as the Endobarrier is intact.
7. PCOS as defined by at least two of the following criteria:

   A. Polycystic ovaries. B. Oligo and/or anovulation C. Clinical (i.e acne, hirsutism) and/or biochemical signs of hyperandrogenism (i.e high levels of Testosterone, Androstendione, 17-hydroxyprogesterone, DHEA-S) and exclusion of other etiologies (congenital adrenal hyperplasia androgen-secreting tumors, Cushing's syndrome).
8. IGT as defined by: the ratio of fasting glucose to fasting insulin <4.5, and/or 2-hour glucose level after a 75-g oral glucose tolerance test between 140-199 mg/dL.
9. Documented FSH levels below 12 IU/L, from any source taken no longer than 3 months before screening.

Exclusion Criteria:

1. Subjects taking systemic corticosteroids or drugs known to affect GI motility within 30 days prior to randomization
2. Subjects receiving any prescription or over the counter weight loss medication within 30 days prior to the Endobarrier insertion procedure (including GLP-1 analogs).
3. Known Diabetes as defined by: fasting plasma glucose ≥126 mg/dL or any plasma glucose ≥200 mg/dL or HbA1c level ≥6.5% .
4. Previous GI surgery that could preclude the ability to place the EndoBarrier device, liner or affect the function of the implant
5. Subjects with a history of abnormal GI anatomical findings documented on imaging study, which in the opinion of the Investigator, may impair implantation of the EndoBarrier device
6. Subjects with active GERD not taking a Proton Pump Inhibitor (PPI), which in the investigator's opinion might interfere with the Endobarrier.
7. Subjects with symptomatic kidney stones within 6 months prior to randomization.
8. Known abnormal pathologies or conditions of the gastrointestinal tract, including ulcers or Crohn's disease, atresias or stenoses, upper gastro-intestinal bleeding conditions
9. Subjects with symptomatic gallstones within 6 months prior to randomization
10. Coagulopathy defined as hgb <10g/dl and platelet < 100,000/ml or diagnosis of hemophilia, factor X deficiencies or fibrinogen abnormalities
11. Any documented history of acute or chronic pancreatitis
12. Subjects requiring prescription antithrombotic therapy (i.e. anticoagulant or antiplatelet agent)
13. Subjects unable to discontinue Aspirin or any other NSAIDs (non-steroidal anti-inflammatory drugs) or any other drugs with bleeding as a potential side effect (i.e coumadin) during the study duration
14. Known diagnosis of systemic lupus erythematosus, scleroderma or other autoimmune connective tissue disorder
15. Subject is or has been enrolled in another investigational study within 3 months of participation into the EndoBarrier study
16. Subjects with poor dentition who cannot completely chew their food.
17. Subjects with thyroid disease unless controlled with a therapeutic dose of medication and have normal thyroid function tests for a minimum of 6 months prior to randomization
18. Subjects not residing within a 3 hour driving distance of the study center.
19. Subjects with an abnormal laboratory or ECG abnormality which the investigators deems clinically significant and makes the patient a poor candidate for the study
20. Subjects with known allergies or hypersensitivity to ceftrixone, cephalosporins or penicillin.
21. The investigator may decide to exclude the participation of a subject due to medical, safety or any other reason (i.e; behavioral issues, etc.) at any point before the implantation procedure.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2014-09; Primary Completion 2017-09 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
change in egg quality or ovulation rate after Endobarrier treatment | 2.5 years
  Different fertility parameters will be tested during IVF treatment after endobarrier treatment: Total number of retrieved oocytes, Number of oocytes in M2, Number of 2PN, Top quality embryos on day of transfer, Number of embryos transferred Number of follicles above 15 mm,E2 on day of HCG, Number of embryos frozen. Ovulation in response to Clomiphene citrate will also be assessed.

SECONDARY OUTCOMES:
percent change in LDL cholesterol | 6 months
percent change in HDL cholesterol | 6 months
percent change in Triglycerides | 6 months
percent change in HbA1c | 6 months
percent change in fasting plasma glucose levels | 6 months
percent change in body mass index | 6 months
percent change in waist circumference | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Gabriella Lieberman, MD, Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel